CLINICAL TRIAL: NCT01478230
Title: A Proof of Concept With a New Nicotine Inhaler in Comparison With Nicotine Inhaler 10 mg
Brief Title: An Exploratory Study Comparing Two Nicotine Inhalers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NICTDP0002; 2011-002796-41 (EudraCT Number)
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N1/3-I5 (Experimental): 5 mg Inhalation during 10 minutes every hour for 11 hours with a puff frequency of four puffs per minute, with a 36-hour washout between visits
  Interventions: Drug: Nicotine
- NX-I10 (Active Comparator): 10 mg Inhalation during 10 minutes every hour for 11 hours with a puff frequency of four puffs per minute, with a 36-hour washout between visits.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Nicotine 5 mg Inhaler
  Other Names: Not yet marketed
  Arms: N1/3-I5
Drug: Nicotine — Nicotine 10 mg Inhaler
  Other Names: Not yet marketed
  Arms: NX-I10

SUMMARY:
Subjects will be screened within 28 days before the first study treatment to confirm that they meet the requirements to participate in the trial. They will return to the site for two treatment visits, at least 12 hours each, and at least one day in between visits. At each visit treatment N1/3-I5 or Nicotine Inhaler 10 mg will be administered every hour for 11 hours. The investigator (or an appropriate delegate at the investigator site) will obtain informed consent from each subject. Blood samples will be drawn on a special schedule. The total predicted amount of blood sampled from each subject is 174 mL over the whole study. Subjects will be required to follow specific smoking and dietary restrictions and rate their urges to smoke, general liking of the product, and how easy the product is to use.

DETAILED DESCRIPTION:
Blood for pharmacokinetic analyses will be drawn prior to the first administration and immediately before administration at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, and 11 hours. Thereafter samples will be drawn at 5, 10, 15, 20, 25, 30, 45, and 60 minutes after the 11-hour administration. Easiness of use will be rated using an 8-grade ordered category scale at 10 minutes after the start of administrations at 3, 6, and 9 hours. Overall liking will be rated using an 8-grade ordered category scale at 12 hours. Urges to smoke will be rated on a 4-grade ordered category scale immediately before and at 15 minutes after the first administration, and as well as before and 15 minutes after the start of administrations at 3, 6, and 9 hours, and at 12 hours. Used cartridges will be collected. Pooled samples per subject and treatment will be analyzed to determine the amount of remaining nicotine. Tolerability of the treatments will be evaluated in terms of reported and observed adverse events (AE).

Since the primary objective is to compare steady-state nicotine pharmacokinetics of N1/3-I5 with that of Nicotine Inhaler 10 mg, this study will have a multiple-dose setting. A crossover design has been chosen for this study in order to allow within-subject comparisons of treatments. Healthy habituated adults smoking at least 10 cigarettes daily for at least one year preceding inclusion will be included in the study, since they are expected to tolerate the doses of nicotine that will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (per protocol-specified parameters) male or female subjects between the ages of 19 and 50 years, inclusive.
* Smoking of at least 10 cigarettes daily during at least one year preceding inclusion.
* For females: Postmenopausal state or premenopausal/perimenopausal state with a protocol-specified effective means of contraception or declared absence of sexual contact with a male partner during the study.
* For males: No pregnant spouse or partner at screening and willingness to protect potential spouse or partner from becoming pregnant during the study.
* Body Mass Index (BMI) within protocol-specified parameters.
* A personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures specified in the protocol

Exclusion Criteria:

* Evidence or history of an acute or chronic medical or psychiatric condition or allergy or laboratory abnormality, or of use of drugs that, in the judgment of the investigator or an authorized study physician, may increase the risk associated with study participation or interfere with the interpretability of study results.
* Females: Pregnancy, breast-feeding, premenopausal, or perimenopausal, state with insufficient contraception as specified under Inclusion Criteria.
* Males: Pregnant spouse or partner or no willingness to prevent conception in a spouse or partner.
* History of regular alcohol consumption outside the protocol-specified allowances.
* Treatment with an investigational drug within 3 months preceding the first dose of study treatment.
* Known sensitivity to heparin or history of heparin-induced thrombocytopenia.
* Pathological oral status interfering with normal muscular, sensory, or absorptive function of the oral cavity. Piercing of tongue and lips is considered to impair oral function.
* Relationship to persons involved directly with the conduct of the study, or their families.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | During last dosing interval 11-12 hours post-dose
  Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, measured in nanograms/milliliter (ng/mL)
Average Concentration (Cav) | During last dosing interval 11-12 hours post-dose
  The average concentration of nicotine in the blood.
  * The dosing interval (τ) in this study will be one (1) hour. Consequently, Cav will have the same value as AUCτ (but with a different unit), since Cav is calculated as AUCτ divided by τ. Therefore Cav will not be displayed in results, only AUCτ.
Bioavailability [AUCτ] | During last dosing interval 11-12 hours post-dose
  AUCτ is the area under the plasma concentration-vs.-time curve during the last dosing interval and is a measure of how much of the drug reaches the person's bloodstream. The Area Under the Curve (AUC) is calculated by plotting the drug's blood levels on a graph at different times during the set period. The area under this curve is calculated as hour * nanograms (ng) per milliliter (mL).

SECONDARY OUTCOMES:
Minimum Observed Plasma Concentration (Cmin) | During last dosing interval 11-12 hours post-dose
  Minimum Observed Plasma Concentration (Cmin), which is the minimum concentration (amount of drug) measurable in blood plasma after a dose is administered, measured in nanograms/milliliter (ng/mL)
Time of Maximum Concentration (Tmax) | During last dosing interval 11-12 hours post-dose
  The time at which maximum concentration is reached (Tmax)
Peak Trough Fluctuation (PTF) | During last dosing interval 11-12 hours post-dose
  Peak trough fluctuation within one dosing interval at steady state.
Swing | During last dosing interval 11-12 hours post-dose
  Swing within one dosing interval at steady state.
Baseline-corrected Pre-Dosing Plasma Concentration (Cn) | 0 Minutes
  Baseline-corrected nicotine plasma concentrations immediately before each user session (Cn)
Residual Nicotine | 12 hours
  Used cartridges will be collected. Pooled samples per subject and treatment will be analyzed to determine the amount of remaining nicotine.
Urges to Smoke | During 12 hours
  Subjects will rate their urges to smoke on a category scale from 1 to 4, where 1= No or very light urge to smoke, and 4= Very strong or extreme urge to smoke.
Overall Liking | at 12 hours
  Overall Liking will be rated on a category scale from 1 to 8, where 1= extremely good and 8=extremely bad.
Ease of Use | During 9 hours
  Ease of use will be rated at specific categorical time points, on a scale of 1-8, where 1= extremely easy and 8=extremely hard..

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- McNeil AB Clinical Pharmacology R&D, Lund, Sweden